CLINICAL TRIAL: NCT06904911
Title: Intra-Arterial Tenecteplase to Improve the Microvascular Hemodynamics After Mechanical Thrombectomy
Acronym: INTIMA-MT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTIMA-MT
Record Dates: First submitted 2025-03-17; First posted 2025-04-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke From Large Vessel Occlusion
Keywords: acute ischemic stroke; ischemic stroke; large vessel occlusion; reperfusion; adjuvant thrombolysis; intra-arterial thrombolysis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- intra-arterial tenecteplase (Experimental): Patients will receive a single dose of tenecteplase, administered intra-arterially after successful large vessel recanalization. The treatment will be administered via intra-arterial catheter in the distal M1 segment of the middle cerebral artery (distal to lenticulostriates).
  Interventions: Drug: intra-arterial tenecteplase administration

INTERVENTIONS:
Drug: intra-arterial tenecteplase administration — Patients will receive a single dose of tenecteplase, administered intra-arterially after successful large vessel recanalization. The treatment will be administered via intra-arterial catheter in the distal M1 segment of the middle cerebral artery (distal to lenticulostriates).
  Other Names: intra-arterial thrombolysis

SUMMARY:
This is a prospective, single-arm, open-label study to evaluate the efficacy of intra-arterial tenecteplase in improving microvascular reperfusion following successful large vessel recanalization. Acute ischemic stroke patients with large anterior circulation large vessel occlusion will receive a single weight-based dose of intra-arterial tenecteplase after achieving successful large vessel recanalization (defined as TICI ≥ 2b) via standard of care mechanical thrombectomy. Microvascular flow will be assessed by quantitative angiography before and after the intra-arterial drug administration in order to quantify the impact of targeted thrombolysis on microvascular reperfusion. Reperfusion will be secondarily assessed with 24-hour imaging, final infarct volume will be quantified 72 hours following treatment, and functional outcome will be assessed in the short-term by the NIHSS and in the long-term by the 90-day modified Rankin Scale.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label pilot trial to evaluate the efficacy of IA-TNK in improving microvascular reperfusion following successful large vessel recanalization. Acute ischemic stroke patients will receive IA-TNK after achieving mTICI ≥ 2b recanalization via standard of care mechanical thrombectomy (MT). Microvascular flow will be assessed by quantitative angiography before and after IA-TNK to quantify the impact of targeted thrombolysis on microvascular reperfusion. Reperfusion will be secondarily assessed with 24-hour imaging. Final infarct volume will be quantified 72 hours following treatment. Functional outcome will be assessed in the short-term by the NIHSS and at 90-days by the modified Rankin Scale.

N=20 acute stroke patients will be enrolled after successful recanalization of a proximal anterior circulation LVO (internal carotid artery or first segment of the middle cerebral artery). After standard of care MT, every patient will undergo a quantitative angiographic assessment with syngo iFLOW (Siemens Healthineers). More specifically, 2D angiographic images will be acquired with a 8 Fr catheter located in the extracranial C2-C4 segment of the internal carotid artery. 6 mLs of contrast agent will be injected at a flow rate of 4 mL/sec (standardized injection via power injector). The 2D imaging will be acquired at a rate of 4 frames per second to acquire images in anterior-posterior and lateral positions. Images will be transferred to the workstation at which syngo iFLOW software will enable quantification of the microvascular cerebral circulation time (mCCT). Post-processing via iFLOW requires 1-2 minutes. ROI selection to quantify mCCT requires approximately 2-5 minutes.

After post-MT mCCT is quantified, the catheter will be advanced to the distal M1 segment of the MCA (distal to lenticulostriates). 0.125 mg/kg (max 12.5mg) of TNK (i.e. 50% of the IV dose) will be administered via a 5-minute intraarterial infusion (using a programmable syringe pump). As described in section 3.3.1, the dose may be modified as clinical trial data become available, if the available data identify an alternative dose to be optimal.

10 minutes post-TNK, the quantitative angiographic assessment will be repeated to calculate the post-treatment mCCT. The primary objective of this trial is to quantify the change in mCCT associated with IA-TNK treatment.

Post-treatment clinical monitoring will continue as per institutional standard of care (post-MT and post-TNK monitoring). Standard of care NCCT, in addition to protocol CTA/CTP, will be performed 24 hours post-TNK to secondarily assess recanalization, reperfusion, and safety (i.e. hemorrhagic complications). Study protocol MRI of the brain will also be performed 72 hours post-TNK to quantify final infarct volume. Serial NIHSS will assess early functional outcome. Dramatic clinical recovery (DCR) will be defined as a ≥8 point improvement in NIHSS between baseline and 24 hours post-TNK. 90-day mRS will assess long-term functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient/legally authorized representative has signed the Informed Consent Form
* At least 18 years of age
* Ability to comply with the study protocol, in the investigator's judgment
* Acute ischemic stroke attributed to anterior circulation large vessel occlusion (of the internal carotid artery or first segment of the middle cerebral artery based on CTA, MRA, or catheter angiogram) being treated with mechanical thrombectomy
* NIHSS ≥ 6 at the initiation of endovascular therapy (arterial puncture)
* Time from stroke onset to IA-TNK administration < 24 hours. Stroke onset is defined as the time the patient was last known to be at their neurologic baseline
* ASPECTS ≥ 6 on pre-MT CT imaging
* If treated > 6 hours from stroke onset, CTP imaging must demonstrates favorable mismatch profile (based on RAPID processing: infarct core <70 mL, mismatch ratio ≥ 1.8 and mismatch volume ≥ 15 mL)
* Qualifying neuroimaging (CT and CTP, if applicable) must be obtained <120 minutes prior to arterial puncture.

Exclusion Criteria:

* Current participation in another investigational drug or device study
* Known hypersensitivity or allergy to any ingredients of tenecteplase
* Active internal bleeding
* Known bleeding diathesis (Alzheimer's patients taking lecanemab)
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; recent oral anticoagulant therapy with INR > 1.7
* Use of one of the new oral anticoagulants within the last 48 hours (dabigatran, rivaroxaban, apixaban, edoxaban)
* Treatment with a thrombolytic within the last 3 months prior to randomization, inclusive of intravenous thrombolysis during the index stroke.
* Baseline platelet count < 100,000/microliter (results must be available prior to treatment)
* Baseline blood glucose > 400 mg/dL (22.20 mmol/L)
* Baseline blood glucose < 50 mg/dL needs to be normalized prior to randomization
* Intracranial or intraspinal surgery or trauma within 2 months
* Other serious, advanced, or terminal illness (investigator's judgment) or life expectancy is less than 6 months
* History of acute ischemic stroke in the last 90 days
* History of hemorrhagic stroke
* Presumed septic embolus; suspicion of bacterial endocarditis
* Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the patient if an endovascular procedure was to be performed
* Pregnant
* Systolic BP >185 mmHg or diastolic BP >110 mmHg, refractory to treatment
* Suspicion of aortic dissection
* Known allergy to iodine or iodinated contrast
* Subject who requires hemodialysis or peritoneal dialysis, or who have a contraindication to an angiogram
* Renal failure as defined by a serum creatinine > 3.0 mg/dl or GFR < 30
* Known intracranial neoplasm
* GI bleeding within the past 21 days
* Pre-existing medical or neurological disease that will confound the neurological or functional evaluations
* Premorbid (prior to the index stroke) modified Rankin Scale (mRS) score ≥ 3

Additional neuroimaging exclusion criteria:

* ASPECTS <6 on pre-MT CT imaging
* Acute intracranial hemorrhage or contrast extravasation on CT before or immediately after MT (prior to study drug administration)
* Significant mass effect with midline shift on non-contrast CT before or immediately after MT
* Cervical or intracranial stent placement during endovascular therapy
* Acute symptomatic arterial occlusions in more than one vascular territory confirmed on CTA, MRA, or catheter angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in microvascular cerebral circulation time (mCCT) | The change in mCCT will be calculated as mCCT immediately preceding intra-arterial tenecteplase minus the mCCT immediately following intra-arterial tenecteplase
  mCCT will be assessed by quantitative angiography, calculated as the difference between the time-to-peak of the Rolandic artery and Rolandic vein.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Favilla, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided